CLINICAL TRIAL: NCT01120288
Title: A Pilot Study of EZN-2968, an Antisense Oligonucleotide Inhibitor of HIF-1alpha, in Adults With Advance Solid Tumors
Brief Title: A Pilot Study of EZN-2968, an Antisense Oligonucleotide Inhibitor of HIF-1alpha, in Adults With Advanced Solid Tumors With Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100113; 10-C-0113
Record Dates: First submitted 2010-05-07; First posted 2010-05-10 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2014-03-06

CONDITIONS: Neoplasms; Liver Metastases
Keywords: Anti-Angiogenesis; Targeted Therapy; HIF; Antisense; VEGF; Cancer; Solid Tumor; Liver Metastasis
MeSH Terms: conditions — Neoplasms | interventions — EZN 2968

INTERVENTIONS:
Drug: EZN-2968

SUMMARY:
Background:

- A protein called HIF is believed to be involved both in forming cancers and helping them to grow after they are formed. EZN-2968 is a new type of cancer drug that goes into the cancer cell and switches off the production of the HIF protein. Researchers are interested in testing EZN-2968 in people who have liver cancer because studies have shown that this drug travels to the liver and stays there when the drug is given through a vein.

Objectives:

- To determine the safety and effectiveness of EZN-2968 on liver cancer.

Eligibility:

- Individuals 18 years of age and older who have been diagnosed with liver cancer that has not responded to standard treatments.

Design:

* Participants will have an initial screening visit with a physical examination, blood and urine tests, and imaging studies to assess tumor size. Tumor biopsies may also be taken for research purposes.
* Participants will have an undefined number of 6-week treatment cycles of EZN-2968, given once a week for 3 weeks followed by 3 weeks without the drug.
* During each cycle, participants will have additional blood tests and imaging scans to assess tumor response to treatment.
* Cycles of treatment with EZN-2968 may continue until the treatment is not effective, illness requires participants to stop taking the study drug, or the participant chooses to withdraw from the study.

DETAILED DESCRIPTION:
Background:

* Hypoxia-inducible factor-1 (HIF-1) facilitates the adaptation of normal and tumor tissue to oxygen deprivation. HIF-1 is frequently overexpressed in cancer cells, where it is involved in the upregulation of many gene products essential for invasion, migration, angiogenesis, and survival, including vascular endothelial growth factor (VEGF). Blocking HIF-1 activity inhibits the expression of VEGF, resulting in the inhibition of tumor growth in vitro and in vivo.
* EZN-2968 is an antisense oligonucleotide that specifically targets HIF-1 alpha, one of the subunits of HIF-1. Safety and preliminary suggestion of activity have been demonstrated in two Phase I trials; one patient with hepatocellular carcinoma, one with renal cell cancer, and one with angiosarcoma of the face treated with EZN-2968 had objective evidence of shrinkage of large masses. In vivo data show evidence of intracellular uptake of EZN-2968 into tumor cells, and in the Phase I trial, preliminary data show that eleven patients had prolonged stable disease (>90 days duration on study), three of which had objective evidence of tumor shrinkage, thus demonstrating proof of principle for this approach.

Primary Objective:

- Determine the modulation of HIF-1alpha mRNA in tumor biopsies pre- and post-administration of EZN-2968.

Secondary Objectives:

* Assess the safety of EZN-2968 in patients with advanced solid tumors.
* Determine the modulation of HIF-1 alpha protein levels in tumor biopsies pre- and post-administration of EZN-2968.
* Evaluate anti-tumor response as determined by RECIST.
* Evaluate the expression of HIF-1 alpha target genes by real-time PCR in tumor biopsies.
* Assess tumor angiogenesis using DCE-MRI.

Eligibility:

* Adult patients with histologically or cytologically confirmed solid malignancies will be included in the study.
* Patients must have disease that is not amenable to potentially curative resection.
* Patients must have failed at least one line of prior therapy for metastatic disease or have a disease for which no standard curative therapy exists.
* Lesion must be amenable to biopsy.

Design:

* EZN-2968 will be administered as a 2-hour IV infusion at a dose of 18 mg/kg once a week for 3 consecutive weeks followed by a 3-week period without drug. Each cycle will be 6 weeks, i.e., 3 weeks of therapy followed by 3 weeks without drug.
* Tumor biopsies and other correlative imaging and pharmacodynamic studies will be performed at baseline and after the third dose. Tumor restaging will be performed every 2 cycles.

ELIGIBILITY:
* Eligibility Criteria

Inclusion Criteria

* Patients must have histologically or cytologically confirmed diagnosis of solid tumor. The diagnosis should be confirmed by the Laboratory of Pathology, NIH.
* Patients must have disease that is not amenable to potentially curative resection.
* Disease must be amenable to biopsy, and patients must be willing to undergo tumor biopsies.
* Patients must have failed at least one line of prior therapy for metastatic disease or have a disease for which no standard curative therapy exists. Prior anti-angiogenic therapy is allowed.
* Age (Bullet)18 years. Because no dosing or adverse event data are currently available on the use of EZN-2968 in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable.
* Life expectancy of greater than 3 months.
* ECOG performance status 0-2 (Karnofsky (Bullet)60%).
* Patients must have normal organ and marrow function as defined below:

absolute neutrophil count (Bullet)1,500/mcL

platelets (Bullet)100,000/mcL

total bilirubin 1.5 X ULN

AST/ALT 2.5 X institutional ULN

creatinine less than or equal to 1.5 x upper limit of normal

OR

creatinine clearance (measured) greater than or equal to 60 mL/minute for patients with creatinine levels >1.5 times upper limit of normal

INR 1.4

PTT 40 seconds unless due to lupus anticoagulant

* Urine protein should be screened by urine analysis for urine protein:creatinine (UPC) ratio. For UPC ratio >1, 24-hour urine protein should be obtained and the level should be <500 mg for patient enrollment.
* The effects of EZN-2968 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (abstinence; female use of hormonal methods, or barrier methods of birth control; male use of a condom) prior to study entry, for the duration of study participation, and for 6 months after completion of study. Because there is a risk for adverse events in nursing infants secondary to treatment of the mother with EZN- 2968, breastfeeding should be discontinued while the patient is on this trial and for

  30 days after completion of treatment on this trial. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Willingness to undergo tumor biopsies for research purposes.

Exclusion Criteria

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events to eligibility levels (by performance status and laboratory criteria outlined above) due to agents administered more than 4 weeks earlier. Patients may have received investigational agent(s) as part of a Phase 0 study (also referred to as an early Phase I study or pre-Phase I study where a sub-therapeutic dose of drug is administered) at the PI's discretion, up to 2 weeks prior to study entry.
* Patients may not be receiving any other investigational agents.
* Patients with active brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients whose brain metastatic disease status remains stable for (Bullet) 3 months after treatment of the brain metastases without steroids or antiseizure medications may be enrolled at the discretion of the principal investigator.
* Patients requiring therapeutic anticoagulation.
* Hypertension not controlled by medical therapy (hypertension defined as systolic blood pressure >150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to EZN-2968.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. A history of hepatitis is allowed if, following consultation with Liver Diseases Branch, it is felt to be clinically stable.
* Pregnant women are excluded from this study because EZN-2968 has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with EZN-2968, breastfeeding should be discontinued if the mother is treated with EZN-2968.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with EZN-2968.
* Patients with surgical non-healing wounds. Patients with other non-healing wounds will be evaluated and included at the PI s discretion if considered minor.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-04-29; Study Completion 2013-09-24 (Actual)

PRIMARY OUTCOMES:
Determine the modulation of HIF-1 alpha mRNA in tumor biopsies pre- and post- administration of EZN-2968. | 1-2 years

SECONDARY OUTCOMES:
Assess the safety of EZN-2968 in patients with liver-predominant solid tumors. Determine the modulation of HIF-1 alpha protein levels in tumor biopsies pre- and post-administration of EZN-2968. | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wenger RH, Rolfs A, Marti HH, Guenet JL, Gassmann M. Nucleotide sequence, chromosomal assignment and mRNA expression of mouse hypoxia-inducible factor-1 alpha. Biochem Biophys Res Commun. 1996 Jun 5;223(1):54-9. doi: 10.1006/bbrc.1996.0845. PMID 8660378
- [Background] Semenza GL. HIF-1 and mechanisms of hypoxia sensing. Curr Opin Cell Biol. 2001 Apr;13(2):167-71. doi: 10.1016/s0955-0674(00)00194-0. PMID 11248550
- [Background] Semenza GL. Targeting HIF-1 for cancer therapy. Nat Rev Cancer. 2003 Oct;3(10):721-32. doi: 10.1038/nrc1187. PMID 13130303